CLINICAL TRIAL: NCT06069323
Title: Therapeutic Use of Repetitive Transcranial Magnetic Stimulation (rTMS) in Pediatric Autism Spectrum Disorder (ASD) and Attention Deficit Hyperactivity Cohorts (ADHD): a Randomized, Sham-controlled Study.
Brief Title: Therapeutic Use of rTMS in Pediatric ASD and ADHD Cohorts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedali Riuniti di Foggia (Other)
Responsible Party: Principal Investigator, Rosa Savino, Principal Investigator, Ospedali Riuniti di Foggia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 50/CE/2023
Record Dates: First submitted 2023-08-30; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Autism Spectrum Disorder; ADHD; Neurodevelopmental Disorders
Keywords: TMS; NEUROMODULATION; ASD; ADHD; NEUROSTIMULATION; COGNITION; EXECUTIVE FUNCTIONS; DLPFC
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: A double-blind randomized, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active ASD group (Active Comparator): The rTMS will be administered 18 times, twice per week, with the following stimulation parameters: 1.0 Hz frequency, 90% MT, 180 pulses per session with 9 trains of 20 pulses each with 20-30s intervals between the trains.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Sham ASD group (Sham Comparator): 18 rTMS sessions will be administered, placing the coil perpendicular to the scalp of the stimulation site, to avoid stimulation.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Active ADHD group (Active Comparator): The rTMS will be administered 18 times, twice per week, with the following parameters: 5-10 Hz frequency, 90% MT, 180 pulses per session with 9 trains of 20 pulses each with 20-30 s intervals between the trains.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Sham ADHD group (Sham Comparator): 18 rTMS sessions will be administered, placing the coil perpendicular to the scalp of the stimulation site, to avoid stimulation.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — Pediatric patients with ASD and ADHD will be randomized both in active and sham groups.
  Other Names: rTMS, Neurostimulation, Neuromodulation

SUMMARY:
In this interventional, pilot clinical trial investigators will stimulate the dorsolateral prefrontal cortex (DLPFC) in patients with Autism and ADHD. The goal of the study is to improve Cognition and Executive Functions associated with this brain region and, consequently, ameliorate the core symptoms of the disorders.

Specifically, the primary purpose is to establish the efficacy, safety, and tolerability of TMS in pediatric patients with ASD and ADHD. Concurrently, the research aims to uncover the impact of TMS on particular biomarkers associated with the development of these disorders and validate the hypothesis suggesting that the BDNF gene polymorphism (Val66Met) could influence an individual's susceptibility to TMS.

Participants will be randomized into the active group and placebo group, to guarantee a real assessment of the impact of neurostimulation on the cognitive, behavioral, and biochemical parameters. Participants will be asked to complete a neuropsychological evaluation and a biological sample collection before and after TMS treatment, and 1-month post-treatment completion.

DETAILED DESCRIPTION:
BACKGROUND ASD and ADHD are complex neurodevelopmental disorders with increasing prevalence worldwide. The neurobiology of ASD and ADHD reveals a complex picture of altered excitation-inhibition (E/I) balance, aberrant neuronal activity, and disorganization of brain networks. While cognitive and behavioral abnormalities in ASD are related to excessive excitability (due to altered cortex cytoarchitecture), especially at the prefrontal lobes, ADHD patients show reduced activation in the right VLPFC and DLPFC. Neuroinflammation, glutamate imbalance, and kynurenines pathway (KP) dysfunction seem to play a key role in the pathogenesis of these disorders, creating a self-sustaining auto-toxic loop. Treatment options for these disorders are limited, mainly focusing on early behavioral interventions. While for ASD there are no specific pharmacological treatments to address the core symptoms, psychostimulants are considered the most effective therapy for patients with ADHD. Unfortunately, various side effects and the potential for abuse with no reduction in symptom severity in long-term use can restrict its administration. In this scenario, transcranial magnetic stimulation (TMS) could emerge as a reliable therapeutic option. TMS involves magnetic stimulation of the brain to cause long-term changes in excitability and neurochemical activity, healing the key neurobiological alterations described above.

Although shreds of evidence on its potential use in ASD-ADHD treatment, there are still critical challenges that limit its use in clinical practice. One of the big issues is the problem of heterogeneity of the results and the stimulation protocols used in current studies.

Many factors influence the efficacy of TMS, including the stimulation parameters and the functional state of the targeted region during stimulation. Also, the psychotropic drugs taken by enrolled patients may affect TMS outcomes, as they cause long-term changes in synaptic and excitatory balance.

The brain-derived neurotrophic factor (BDNF) gene polymorphism (Val66Met) has been considered a critical contributing factor to individual susceptibility to TMS. BDNF is, indeed involved in early and long-term potentiation, particularly in hippocampal synapses, and its polymorphism has been shown to affect different cognitive functions. According to the most recent data, heterozygous Val/Met individuals were less susceptible to TMS effects.

Finally, another crucial weakness is the lack of longitudinal follow-up, at a well-defined point in time, later neurostimulation. This avoids critical questions regarding possible predictors of outcome (e.g., genetic profiling), length of persistence of benefits, assessing outcome according to the severity of phenotypic presentation, and utility of booster session.

AIMS and OBJECTIVES

The primary aim of the study is to establish the efficacy, safety, and tolerability of TMS in pediatric patients with ASD and ADHD. Key objectives include:

1. Evaluating TMS impact on core symptoms, cognition, and executive functions.
2. Analyzing changes in peripheral biomarkers, such as neurotransmitters, kynurenines, and neurotrophins following TMS.
3. Investigating the role of BDNF gene polymorphism (Val66Met) in TMS individual susceptibility.
4. Identifying clinical profiles and individual factors influencing TMS efficacy (such as cognitive level, ongoing therapies, age, sex, neuropsychiatric comorbidities, clinical severity, etc.).
5. Establishing a longitudinal follow-up to assess predictors of outcome, persistence of benefits, and the utility of booster sessions.

METHODOLOGY It is expected to recruit for this study at least 80 children, divided into 2 groups: 40 children with ASD, and 40 children with ADHD, both of them will be randomly divided into the active group (real TMS stimulation) and the Sham group (placebo stimulation). In case of the inferiority of the sample, due to the difficulty of recruitment, investigators will proceed to administer the active and sham stimulation to the same patients, alternatively, in two different moments, after a proper wash-out. It has been proposed 36-40 months to complete the whole study.

Recruitment of participants will be carried out at the Neuropsychiatry Unit for Children and Adolescents, General Hospital "Riuniti" of Foggia. It has been planned to identify children among hospitalized patients who need a first diagnosis of ADHD and ASD or who need to be followed up. Written informed consent will then be requested from parents, legal tutors, and children wherever possible.

* Study Assessment

This study will be articulated according to the following phases:

1. Collecting and managing biomaterials Peripheral blood, saliva, and urine samples will be collected before and after neurostimulation.

   To verify the impact of TMS on serum and molecular profile in children with neurodevelopmental disorders, we will provide a third biological sample, one month after the last neurostimulation session.

   The following biomarkers will be assessed:

   • Tryptophan and its catabolites: KINA, QUIN, 3-HK, etc.

   • Glutamate, GABA (γ-Aminobutyric acid), Serotonin, and Dopamine.
   * Plasmatic BDNF
   * Inflammatory biomarkers: cortisol, IL-6, IL-1β, TNF-α, TSH, FT3, FT4, Protein-C-reactive (PCR), ferritin.

   A small amount of blood will be used to genotype BDNF gene polymorphism (Val66Met).
2. Clinical and Neuropsychological assessment

   Parents will be asked to complete a set of questionnaires and interview measures designed to assess symptoms of ASD and ADHD, such as:

   • Vineland Adaptive Behavior Scales - Second Edition.

   • Conners 3

   • The Child Behavior Checklist (CBCL).

   • Autism Diagnostic Interview-Revised (ADI-R)

   • Social Communication Questionnaire (SCQ).

   Participants will be asked to complete a battery of cognitive, neuropsychological, and play-based assessments, including:

   • Autism Diagnostic Observation Schedule-2 (ADOS-2).
   * Wechsler Intelligence Scale for Children IV Ed.
   * Leiter International Performance Scale-Revised.
   * Developmental Neuropsychological Assessment, second edition (NEPSY-II)
   * M-ABC (Movement Assessment Battery for Children)
   * Children's Depression Inventory 2™ (CDI 2)
   * Multidimensional Anxiety Scale for Children Second Edition™ (MASC 2)

   Neuropsychological evaluation will be conducted at three different moments, before and after the neurostimulation and 1 month after the last stimulation.
3. EEG data collection and Neurostimulation The Department of Clinical and Experimental Medicine-University of Foggia will perform TMS neurostimulation.

For all participants (both active and sham groups), EEG data will be recorded two times, 30 min before TMS and within 30 min after the last stimulation. The participants will sit in a quiet room, awake and relaxed, with their eyes open. During the data-recording process, 5-10 minutes of resting-state EEG data will be recorded from 32 electrodes positioned according to the 10-10 International System (BrainVision, Brain Products GmbH, Germany).

Matlab and the package EEG lab will be used for offline data analysis.

TMS parameters will be tailored to each disorder's neurobiology. - ASD Protocol The Casanova-Sokhadze research group's TMS protocol will be used because it is the most widely replicated protocol in the pediatric population, with good safety and tolerability as well as fair efficacy.

For repetitive TMS administration, we will use a Magstim R2 stimulator (Magstim Co, UK) with a 70-mm wingspan figure-eight coil, handle oriented approximately 45° from the midline. The neuronavigation system will be utilized to correctly identify the stimulation site (PFC/DLPFC) for every subject. Since it is difficult to treat patients with autism, to avoid their discomfort researchers hypothesize establishing the location of TMS stimulation, through the use of anatomical landmarks corresponding to the scalp regions used for F3 and F4 EEG electrode placement in the 10-20 international system.

Individual MT will be assessed for each hemisphere at the beginning of treatment (L DLPFC, R DLPFC, L + R DLPFC).

Participants will receive 18 rTMS treatment with Fig8 coil twice weekly (9 weeks). The rTMS will be administered with the following stimulation parameters: 1Hz frequency, 90% MT, 180 pulses per session with 9 trains of 20 pulses each with 20-30s intervals between the trains. The initial 6 times, rTMS sessions will be administered over the left DLPFC, followed by 6 sessions targeting the right DLPFC, and an additional 6 treatments will be done bilaterally. The sham rTMS group will receive the same process but the figure-eight coil will be placed vertically on the scalp with no magnetic field penetrated through the skull. The stimulation parameters will be the same as those of the real rTMS. The environmental conditions will be the same for each test (comfortable armchair, quiet room, elbow positioned at 90◦ flexion). Participants will be required to use earplugs during TMS sessions.

The selection of 90% of the Motor Threshold (MT) has been chosen as a precautionary measure to reduce the risk of seizure in this study population, while the choice of 1 Hz of stimulation is based on the evidence that low-frequency improves cortex E/I imbalance.

- ADHD protocol Participants will receive 18 rTMS treatments with Fig-8 coil twice per week (9 weeks). The rTMS will be administered with the following stimulation parameters: 5 (or 10) Hz frequency, 90% MT, 180 pulses per session with 9 trains of 20 pulses each with 20-30 s intervals between the trains. The initial six times, rTMS sessions will be administered over the left DLPFC, followed by 6 sessions targeting the right DLPFC, and an additional 6 treatments will be done bilaterally (over the left and right DLPFC). For the sham rTMS group, the coil will be simply placed perpendicular to the scalp of the stimulation site. The stimulation parameters will be the same as those of the real rTMS.

Studies on children and adolescents with ADHD are significantly fewer than those with ASD. So it is difficult to find a validated and often replicated TMS protocol. For the ADHD population, high-frequency stimulation will be used since it was noted that high frequency can significantly improve ADHD symptoms. It has been also shown that TMS might produce a similar effect on the dopamine system as D-amphetamine a well-known psychostimulant. It has been decided to select 90% of the MT to avoid seizure risk to patients.

At the end of every single session, a questionnaire regarding side effects will be administered to all participants.

BENEFITS AND IMPLICATIONS The study aims to establish a standardized TMS protocol for pediatric ASD and ADHD, addressing heterogeneity in methodology and outcomes.

Since it has been demonstrated that younger age is a predictor of better response to TMS therapy (as children's brains are more plastic than adults), intervening in the pediatric population might result in more effective effects.

Insights into neurotransmitter and biochemical modulation, BDNF's role, and TMS susceptibility can guide personalized interventions. The research could modernize treatment approaches, offering a noninvasive, targeted therapy for these complex disorders. Additionally, the study might identify potential biomarkers for diagnostic and therapeutic purposes.

ETHICAL CONSIDERATIONS AND CONFIDENTIALITY The study has received ethical approval and complies with the Declaration of Helsinki. Personal data will be securely stored, anonymized, and accessible only to authorized personnel. Stringent measures will be taken to ensure participant confidentiality throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received a diagnosis of "ASD" or "ADHD" according to the Diagnostic and Statistical Manual of Mental Disorder-Fifth edition.
* Patients must be older than 6-7 years of age, to obtain their collaboration easily

Exclusion Criteria:

* presence of known neurological or genetic conditions that are known to affect brain function and structure (i.e. brain tumors, X-fragile, tuberous sclerosis, etc.).
* prescription of psychoactive medication(s) less than 4 weeks prior to joining the study.
* medical history of head trauma associated with prolonged loss of consciousness.
* presence of epilepsy, or history of previous epilepsy, seizures, and repeated febrile seizures.
* presence of comorbidity with psychosis disorder.
* presence of known endocrine, cardiovascular, pulmonary, liver, kidney, or other medical diseases.
* vision and auditory impairment.
* presence of diagnosed chronic or acute inflammation and/or infection.
* lack of consent.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Determining the impact of rTMS on Cognitive Functioning in Real Groups versus Sham Groups, through changes in scores of NEPSY-II sub-scales | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  The NEPSY-II is a comprehensive neuropsychological battery for children and adolescents ages 3-16. It contains 32 subtests, which are divided into six domains of cognitive functioning: Attention and Executive Functioning; Language; Memory and Learning; Sensorimotor; Social Perception; and Visuospatial Processing. Scores are categorized into standard scores (which usually range from 1 to 19 for each subtest), percentile ranks, and age-equivalent scores.
  Results are compared to a normative sample to assess a child's performance. Higher scores generally indicate better performance, while lower scores may suggest areas of concern or developmental delay.
Determining the impact of rTMS on Depression in Real Groups vs. Sham Groups, through changes in CDI and MASC scores | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  The CDI is a self-report questionnaire designed to assess depressive symptoms in children and adolescents. Each item is rated on a scale, often from 0 to 2 or 0 to 3, with higher scores indicating more severe depressive symptoms. The total score is calculated by summing the individual item scores. Cutoff scores are used to categorize depression severity (e.g., mild, moderate, severe).
Determining the impact of rTMS on Motor Skills and Coordination in Real Groups vs. Sham Groups, through changes in M-ABC scores | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  The Movement Assessment Battery for Children (M-ABC) is a motor assessment tool for children aged 3 to 16. The test includes various motor tasks grouped into three categories: manual dexterity, aiming and catching, and balance. Trained examiners administer the tasks and assign scores based on the child's performance. Scores are typically assigned on a scale of 0 to 5 for each task, with higher scores indicating better motor performance. The overall score is calculated by summing the individual task scores within each category. Lower overall scores may suggest motor skill difficulties or delays. The M-ABC results are often interpreted in conjunction with the child's age and gender, as motor development can vary among children.
Determining the impact of rTMS on Emotional and Behavioral Problems in Real Groups vs. Sham Groups, through changes in CBCL scores | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  The Child Behavior Checklist (CBCL) is a questionnaire completed by parents or caregivers to assess a child's behavioral and emotional problems. Parents or caregivers provide responses to a series of questions about the child's behavior and emotions. Each item is assigned a numerical value based on the caregiver's responses. These values are summed to create raw scores for different scales and subscales within the CBCL. The raw scores are then converted into T-scores. T-scores are standardized scores with a mean (average) of 50 and a standard deviation of 10. These scores allow for comparisons with a normative sample of children of the same age and gender. Typically, scores falling within the range of 30 to 70 are considered within the average range. Scores below 30 may indicate below-average functioning, while scores above 70 suggest above-average or potentially concerning behavior.
Determining the impact of rTMS on Adaptive Behaviors in Real Groups vs. Sham Groups, through changes in Vineland Scale scores | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  The Vineland is a structured interview with a parent or caregiver, which assesses adaptive behaviors in four main domains: Communication, Daily Living Skills, Socialization, and Motor Skills (optional). The Vineland uses standard scores percentile ranks, and age-equivalent scores to quantify an individual's level of adaptive functioning. Ratings are typically on a scale with options like "unable," "sometimes," "usually," and "always. These scores are based on the person's performance relative to a normative sample of individuals of the same age. The Vineland provides an overall summary score known as the Adaptive Behavior Composite (ABC) score. It represents an individual's general adaptive functioning across all domains. In addition to the ABC score, the Vineland provides subdomain scores for each of the four main domains, allowing for a more detailed assessment of specific areas.
Determining the impact of rTMS on ADHD symptoms in Real Groups vs. Sham Groups, through changes in Conners scores | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  The Conners-3 (Conners 3rd Edition) is a widely used questionnaire for evaluating and measuring ADHD symptoms in children and adolescents. It may be administered to parents, teachers, and sometimes the child or adolescent themselves, depending on their age.
  The Conners-3 generates standard scores for various scales and indices. These scores are typically presented as T-scores, with a mean of 50 and a standard deviation of 10. T-scores help compare the child's behavior to a normative sample of children of the same age and gender. Higher T-scores indicate more severe symptoms or concerns.
Determining the impact of rTMS on Anxiety in Real Groups vs. Sham | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  MASC is a self-report questionnaire designed to assess anxiety symptoms in children and adolescents. Patients rate the frequency of their experiences on a 4-point scale, with higher scores indicating greater anxiety. MASC provides a total anxiety score, reflecting the overall level of anxiety symptoms. Subscale scores may also be considered to examine specific domains of anxiety ( including physical symptoms, harm avoidance, social anxiety, and separation/panic). Higher total scores on MASC indicate more significant anxiety symptoms.

SECONDARY OUTCOMES:
Determining the impact of rTMS on BDNF in Real Groups vs. Sham Groups, through changes in BDNF serum concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  BDNF levels in the plasma will be measured using laboratory techniques such as enzyme-linked immunosorbent assay (ELISA) or immunoassay. These assays use antibodies that specifically bind to BDNF, allowing for quantification. The results of the assay will be analyzed to determine the concentration of BDNF in the plasma sample. This concentration will be reported in picograms per milliliter (pg/mL).
Determining the impact of rTMS on GABA in Real Groups vs. Sham Groups, through changes in serum concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  Neurotransmitter GABA will be dosed in serum at three different points in time (baseline, post-treatment, and 1 month later), to evaluate the effect of rTMS in modulating its concentration. This neurotransmitter will be quantified by HPLC and mass spectrometry. Concentrations will be reported in nanograms per milliliter (ng/mL) or picomoles per milliliter (pmol/mL), depending on the assay's sensitivity.
Determining the impact of rTMS on glutamate in Real Groups vs. Sham Groups, through changes in serum concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  Glutamate will be dosed in serum at three different points in time (baseline, post-treatment, and 1 month later), to evaluate the effect of rTMS in modulating its concentration. This neurotransmitter will be quantified by HPLC and mass spectrometry. Concentrations will be reported in nanograms per milliliter (ng/mL) or picomoles per milliliter (pmol/mL), depending on the assay's sensitivity.
Determining the impact of rTMS on dopamine in Real Groups vs. Sham Groups, through changes in serum concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  Dopamine will be dosed in serum at three different points in time (baseline, post-treatment, and 1 month later), to evaluate the effect of rTMS in modulating its concentration. This neurotransmitter will be quantified by HPLC and mass spectrometry. Concentrations will be reported in nanograms per milliliter (ng/mL) or picomoles per milliliter (pmol/mL), depending on the assay's sensitivity.
Determining the impact of rTMS on serotonin in Real Groups vs. Sham Groups, through changes in serum concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  Serotonin will be dosed in serum at three different points in time (baseline, post-treatment, and 1 month later), to evaluate the effect of rTMS in modulating its concentration. This neurotransmitter will be quantified by HPLC and mass spectrometry. Concentrations will be reported in nanograms per milliliter (ng/mL) or picomoles per milliliter (pmol/mL), depending on the assay's sensitivity.
Determining the impact of rTMS on Kynurenines Pathway in Real Groups vs. Sham Groups, through changes in kynurenines serum and urine concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  Kynurenines will be extracted from urine, saliva, and plasma, at three different points in time (baseline, post-treatment, and 1 month later). The main goal is to evaluate how TMS intervention influences the Kynurenines pathway, involved in neuroinflammation. Kynurenines level will be measured using high-performance liquid chromatography (HPLC) or mass spectrometry. The results of the assay will provide the concentration of kynurenines in the respective samples, reported in micromoles per liter (µmol/L) or picomoles per milliliter (pmol/mL) depending on the assay's sensitivity.
Determining the impact of rTMS on inflammatory protein IL-1 in Real Groups vs. Sham Groups, through changes in serum concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  IL-1 will be assessed in the serum to evaluate if TMS impacts its level, as ASD and ADHD pathogenesis involves neuroinflammation. To measure IL-1 enzyme-linked immunosorbent assay (ELISA) will be performed. Concentrations will be reported in nanograms per milliliter (ng/mL) or picomoles per milliliter (pmol/mL), depending on the assay's sensitivity.
Determining the impact of rTMS on inflammatory protein IL-6 in Real Groups vs. Sham Groups, through changes in serum concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  IL-6 will be assessed in the serum to evaluate if TMS impacts its level, as ASD and ADHD pathogenesis involves neuroinflammation. To measure interleukin enzyme-linked immunosorbent assay (ELISA) will be performed. Concentrations will be reported in nanograms per milliliter (ng/mL) or picomoles per milliliter (pmol/mL), depending on the assay's sensitivity.
Determining the impact of rTMS on inflammatory protein TNF-a in Real Groups vs. Sham Groups, through changes in serum concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  Inflammatory proteins, including TNF-a, will be assessed in the serum to evaluate if TMS impacts its levels, as ASD and ADHD pathogenesis involves neuroinflammation. To measure interleukin enzyme-linked immunosorbent assay (ELISA) will be performed. Concentrations will be reported in nanograms per milliliter (ng/mL) or picomoles per milliliter (pmol/mL), depending on the assay's sensitivity.
Determining the impact of rTMS on inflammatory protein CRP (c-reactive protein) in Real Groups vs. Sham Groups, through changes in serum concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  Inflammatory proteins, including CRP, will be assessed in the serum to evaluate if TMS impacts its levels, as ASD and ADHD pathogenesis involves neuroinflammation. To measure interleukin enzyme-linked immunosorbent assay (ELISA) will be performed. Concentrations will be reported in nanograms per milliliter (ng/mL) or picomoles per milliliter (pmol/mL), depending on the assay's sensitivity.
Determining the impact of rTMS on cortisol in Real Groups vs. Sham Groups, through changes in serum and saliva concentration. | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  Cortisol will be assessed in the serum and saliva at three different points in time. Immunoassays (ELISA) will be used to quantify it. Results will be typically reported in nanograms per milliliter (ng/mL).

OTHER OUTCOMES:
Determining the impact of rTMS on Event-related potentials (ERPs) in Real Groups vs. Sham Groups, and intra-groups | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  ERPs elicited by TMS will be scored by analyzing their latency and amplitude from EEG data collected.
Determining the impact of rTMS on Resting State-EEG in Real Groups vs. Sham Groups, and intra-groups | Baseline; Post rTMS (9 weeks after baseline); One month follow-up (4 weeks after rTMS)
  Fifteen minutes of resting state will be performed. Free epochs will be finally analyzed in terms of Power Spectral Density and Connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Anna N Polito, MD, Study Chair — Neuropsychiatric Unit for Child and Adolescent, at General Hospital "Riuniti" of Foggia
Locations (1):
- Neuropsychiatric Unit for Child and Adolescent, at General Hospital "Riuniti" of Foggia, University of Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in future articles, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Result] Casanova MF, Buxhoeveden D, Gomez J. Disruption in the inhibitory architecture of the cell minicolumn: implications for autism. Neuroscientist. 2003 Dec;9(6):496-507. doi: 10.1177/1073858403253552. PMID 14678582
- [Result] Casanova MF, Sokhadze EM, Casanova EL, Li X. Transcranial Magnetic Stimulation in Autism Spectrum Disorders: Neuropathological Underpinnings and Clinical Correlations. Semin Pediatr Neurol. 2020 Oct;35:100832. doi: 10.1016/j.spen.2020.100832. Epub 2020 Jun 24. PMID 32892959
- [Result] Hart H, Radua J, Nakao T, Mataix-Cols D, Rubia K. Meta-analysis of functional magnetic resonance imaging studies of inhibition and attention in attention-deficit/hyperactivity disorder: exploring task-specific, stimulant medication, and age effects. JAMA Psychiatry. 2013 Feb;70(2):185-98. doi: 10.1001/jamapsychiatry.2013.277. PMID 23247506
- [Result] Norman LJ, Carlisi C, Lukito S, Hart H, Mataix-Cols D, Radua J, Rubia K. Structural and Functional Brain Abnormalities in Attention-Deficit/Hyperactivity Disorder and Obsessive-Compulsive Disorder: A Comparative Meta-analysis. JAMA Psychiatry. 2016 Aug 1;73(8):815-825. doi: 10.1001/jamapsychiatry.2016.0700. PMID 27276220
- [Result] Rubio B, Boes AD, Laganiere S, Rotenberg A, Jeurissen D, Pascual-Leone A. Noninvasive Brain Stimulation in Pediatric Attention-Deficit Hyperactivity Disorder (ADHD): A Review. J Child Neurol. 2016 May;31(6):784-96. doi: 10.1177/0883073815615672. Epub 2015 Dec 10. PMID 26661481
- [Result] Anderson G, Maes M. Interactions of Tryptophan and Its Catabolites With Melatonin and the Alpha 7 Nicotinic Receptor in Central Nervous System and Psychiatric Disorders: Role of the Aryl Hydrocarbon Receptor and Direct Mitochondria Regulation. Int J Tryptophan Res. 2017 Feb 16;10:1178646917691738. doi: 10.1177/1178646917691738. eCollection 2017. PMID 28469467
- [Result] Savino R, Carotenuto M, Polito AN, Di Noia S, Albenzio M, Scarinci A, Ambrosi A, Sessa F, Tartaglia N, Messina G. Analyzing the Potential Biological Determinants of Autism Spectrum Disorder: From Neuroinflammation to the Kynurenine Pathway. Brain Sci. 2020 Sep 11;10(9):631. doi: 10.3390/brainsci10090631. PMID 32932826
- [Result] Lim CK, Essa MM, de Paula Martins R, Lovejoy DB, Bilgin AA, Waly MI, Al-Farsi YM, Al-Sharbati M, Al-Shaffae MA, Guillemin GJ. Altered kynurenine pathway metabolism in autism: Implication for immune-induced glutamatergic activity. Autism Res. 2016 Jun;9(6):621-31. doi: 10.1002/aur.1565. Epub 2015 Oct 24. PMID 26497015
- [Result] Sathappan AV, Luber BM, Lisanby SH. The Dynamic Duo: Combining noninvasive brain stimulation with cognitive interventions. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Mar 8;89:347-360. doi: 10.1016/j.pnpbp.2018.10.006. Epub 2018 Oct 9. PMID 30312634
- [Result] Cortese S. The neurobiology and genetics of Attention-Deficit/Hyperactivity Disorder (ADHD): what every clinician should know. Eur J Paediatr Neurol. 2012 Sep;16(5):422-33. doi: 10.1016/j.ejpn.2012.01.009. Epub 2012 Feb 2. PMID 22306277
- [Result] Cortese S, Holtmann M, Banaschewski T, Buitelaar J, Coghill D, Danckaerts M, Dittmann RW, Graham J, Taylor E, Sergeant J; European ADHD Guidelines Group. Practitioner review: current best practice in the management of adverse events during treatment with ADHD medications in children and adolescents. J Child Psychol Psychiatry. 2013 Mar;54(3):227-46. doi: 10.1111/jcpp.12036. Epub 2013 Jan 7. PMID 23294014
- [Result] Oberman LM, Enticott PG, Casanova MF, Rotenberg A, Pascual-Leone A, McCracken JT; TMS in ASD Consensus Group. Transcranial magnetic stimulation in autism spectrum disorder: Challenges, promise, and roadmap for future research. Autism Res. 2016 Feb;9(2):184-203. doi: 10.1002/aur.1567. Epub 2015 Nov 4. PMID 26536383
- [Result] Oberman LM, Enticott PG. Editorial: The safety and efficacy of noninvasive brain stimulation in development and neurodevelopmental disorders. Front Hum Neurosci. 2015 Oct 2;9:544. doi: 10.3389/fnhum.2015.00544. eCollection 2015. No abstract available. PMID 26483661
- [Result] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Result] Barahona-Correa JB, Velosa A, Chainho A, Lopes R, Oliveira-Maia AJ. Repetitive Transcranial Magnetic Stimulation for Treatment of Autism Spectrum Disorder: A Systematic Review and Meta-Analysis. Front Integr Neurosci. 2018 Jul 9;12:27. doi: 10.3389/fnint.2018.00027. eCollection 2018. PMID 30038561
- [Result] Sasaki R, Kojima S, Onishi H. Do Brain-Derived Neurotrophic Factor Genetic Polymorphisms Modulate the Efficacy of Motor Cortex Plasticity Induced by Non-invasive Brain Stimulation? A Systematic Review. Front Hum Neurosci. 2021 Sep 28;15:742373. doi: 10.3389/fnhum.2021.742373. eCollection 2021. PMID 34650418
- [Result] Egan MF, Kojima M, Callicott JH, Goldberg TE, Kolachana BS, Bertolino A, Zaitsev E, Gold B, Goldman D, Dean M, Lu B, Weinberger DR. The BDNF val66met polymorphism affects activity-dependent secretion of BDNF and human memory and hippocampal function. Cell. 2003 Jan 24;112(2):257-69. doi: 10.1016/s0092-8674(03)00035-7. PMID 12553913
- [Result] Blum R, Konnerth A. Neurotrophin-mediated rapid signaling in the central nervous system: mechanisms and functions. Physiology (Bethesda). 2005 Feb;20:70-8. doi: 10.1152/physiol.00042.2004. PMID 15653842
- [Result] Abellaneda-Perez K, Martin-Trias P, Casse-Perrot C, Vaque-Alcazar L, Lanteaume L, Solana E, Babiloni C, Lizio R, Junque C, Bargallo N, Rossini PM, Micallef J, Truillet R, Charles E, Jouve E, Bordet R, Santamaria J, Rossi S, Pascual-Leone A, Blin O, Richardson J, Jovicich J, Bartres-Faz D. BDNF Val66Met gene polymorphism modulates brain activity following rTMS-induced memory impairment. Sci Rep. 2022 Jan 7;12(1):176. doi: 10.1038/s41598-021-04175-x. PMID 34997117
- [Result] Casanova MF, Sokhadze EM, Casanova EL, Opris I, Abujadi C, Marcolin MA, Li X. Translational Neuroscience in Autism: From Neuropathology to Transcranial Magnetic Stimulation Therapies. Psychiatr Clin North Am. 2020 Jun;43(2):229-248. doi: 10.1016/j.psc.2020.02.004. Epub 2020 Apr 8. PMID 32439019
- [Result] Casanova MF, Shaban M, Ghazal M, El-Baz AS, Casanova EL, Sokhadze EM. Ringing Decay of Gamma Oscillations and Transcranial Magnetic Stimulation Therapy in Autism Spectrum Disorder. Appl Psychophysiol Biofeedback. 2021 Jun;46(2):161-173. doi: 10.1007/s10484-021-09509-z. PMID 33877491
- [Result] Casanova MF, Shaban M, Ghazal M, El-Baz AS, Casanova EL, Opris I, Sokhadze EM. Effects of Transcranial Magnetic Stimulation Therapy on Evoked and Induced Gamma Oscillations in Children with Autism Spectrum Disorder. Brain Sci. 2020 Jul 3;10(7):423. doi: 10.3390/brainsci10070423. PMID 32635201
- [Result] Kang J, Zhang Z, Wan L, Casanova MF, Sokhadze EM, Li X. Effects of 1Hz repetitive transcranial magnetic stimulation on autism with intellectual disability: A pilot study. Comput Biol Med. 2022 Feb;141:105167. doi: 10.1016/j.compbiomed.2021.105167. Epub 2021 Dec 23. PMID 34959111
- [Result] Cardullo S, Gomez Perez LJ, Cuppone D, Sarlo M, Cellini N, Terraneo A, Gallimberti L, Madeo G. A Retrospective Comparative Study in Patients With Cocaine Use Disorder Comorbid With Attention Deficit Hyperactivity Disorder Undergoing an rTMS Protocol Treatment. Front Psychiatry. 2021 Mar 25;12:659527. doi: 10.3389/fpsyt.2021.659527. eCollection 2021. PMID 33841218
- [Result] Jannati A, Oberman LM, Rotenberg A, Pascual-Leone A. Assessing the mechanisms of brain plasticity by transcranial magnetic stimulation. Neuropsychopharmacology. 2023 Jan;48(1):191-208. doi: 10.1038/s41386-022-01453-8. Epub 2022 Oct 5. PMID 36198876
- [Result] Giron CG, Lin TTZ, Kan RLD, Zhang BBB, Yau SY, Kranz GS. Non-Invasive Brain Stimulation Effects on Biomarkers of Tryptophan Metabolism: A Scoping Review and Meta-Analysis. Int J Mol Sci. 2022 Aug 26;23(17):9692. doi: 10.3390/ijms23179692. PMID 36077088
- [Result] Regenold WT, Deng ZD, Lisanby SH. Noninvasive neuromodulation of the prefrontal cortex in mental health disorders. Neuropsychopharmacology. 2022 Jan;47(1):361-372. doi: 10.1038/s41386-021-01094-3. Epub 2021 Jul 16. PMID 34272471
- [Result] Lisanby SH. Transcranial Magnetic Stimulation in Psychiatry: Historical Reflections and Future Directions. Biol Psychiatry. 2024 Mar 15;95(6):488-490. doi: 10.1016/j.biopsych.2023.05.001. Epub 2023 May 9. No abstract available. PMID 37169276
- [Derived] Savino R, Davinelli S, Polito AN, Scapagnini G, Scirano A, Valenzano A, Cibelli G. Repetitive transcranial magnetic stimulation in children and adolescents with autism spectrum disorder: study protocol for a double-blind, sham-controlled, randomized clinical trial. Trials. 2025 Jul 7;26(1):240. doi: 10.1186/s13063-025-08946-z. PMID 40619411